CLINICAL TRIAL: NCT03599869
Title: Management of Mixed-Phenotype Acute Leukemia in the East of France
Acronym: ELABEST
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: PSS2017/ELABEST-BONMATI/VS
Record Dates: First submitted 2018-06-22; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Mixed Phenotype Acute Leukemia
MeSH Terms: conditions — Leukemia, Biphenotypic, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical presentation and management of Mixed-Phenotype Acute leukemia (MPAL) is heterogeneous. This descriptive observationnal study aims to review MPAL cases in the East of France based on a 10-year multicentre retrospective collection.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over 18 years of age
* Diagnosis of biphenotypic acute leukemia or mixed-phenotype acute leukemia between 2008 and 2018

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients from one of the following 7 hospitals : Nancy, Metz-Thionville, Reims, Strasbourg, Mulhouse, Dijon, Besançon
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Age of the patients when diagnosed with MPAL | At inclusion (Day 0)
  Age in years
Sex of the patients when diagnosed with MPAL | At inclusion (Day 0)
  Male or female
City of the hematology unit in charge of each patient for the treatment of MPAL | At inclusion (Day 0)
  Nancy, Metz-Thionville, Reims, Strasbourg, Mulhouse, Dijon or Besançon
MPAL rate in the each hematology unit | 10 years (01/01/2008-01/01/2018)
  Rate of MPAL out of the total number of patients diagnosed with acute leukemia in each hematology unit
Date of MPAL diagnosis for each patient | At inclusion (Day 0)
Type of MPAL for each patient | At inclusion (Day 0)
  De novo MPAL or secondary to myelodysplasia MPAL
Percentage of blood blasts for each patient at diagnosis of MPAL | At inclusion (D0)
  On the first blood sample analyzed
Percentage of medullar blasts for each patient at diagnosis of MPAL | At inclusion (Day 0)
  On the first bone marrow sample analyzed
Cytologic characteristics: type of myeloid markers at diagnosis for each patient | At inclusion (Day 0)
  Presence or not of myeloid markers generally sought in the diagnosis of acute leukaemias
Cytologic characteristics: type of B lymphoid markers at diagnosis for each patient | At inclusion (Day 0)
  Presence or not of B lymphoid markers generally sought in the diagnosis of acute leukaemias
Cytologic characteristics: type of T lymphoid markers | At inclusion (D0)
  Presence or not of T lymphoid markers generally sought in the diagnosis of acute leukemias
Medullar MPO positivity percentage at diagnosis for each patient | At inclusion (Day 0)
  If performed on the bone marrow sample used to confirm the diagnosis
Genetic characteristics on the caryotype at diagnosis for each patient | At inclusion (Day 0)
  Presence or not of caryotypic abnormalities generally sought in the diagnosis of acute leukemias
Genetic characteristics on molecular biology analysis at diagnosis for each patient | At inclusion (D0)
  Presence or not of molecular biology abnormalities generally sought in the diagnosis of acute leukemias
Classification of biphenotypic acute leukemia (BAL) according to the EGIL 1998 criterias at diagnosis | At inclusion (Day 0)
  BAL or not
Classification of MPAL according to the WHO 2008 criterias at diagnosis | At inclusion (Day 0)
  MPAL or not
Type of treatments and dates of the first day of every treatment line for each patient | 10 years (01/01/2008-01/01/2018)
  Myeloid or lymphoid chemotherapy regimen
Medullar response for every treatments line for each patient | 10 years (01/01/2008-01/01/2018)
  Complete cytological and molecular response or treatment failure
Treatment including allogenic hematopoietic stem cells transplant (HSCT) (yes or no) with type of conditionning regimen for each patient | 10 years (01/01/2008-01/01/2018)
  High-dose, reduced-intensity or nonmyeloablative conditioning regimens with or without total body irradiation
HSCT complicated with acute and/or chronic graft-versus-host disease with severity grade and treatments for each patient | 10 years (01/01/2008-01/01/2018)
  Diagnosis of GVHD according to Filipovich criterias (BMT 2005); Severity grade according to Seattle criterias; Type of treatments: steroids, other immunosuppressive agents, extracorporeal photopheresis

SECONDARY OUTCOMES:
Date of every relapse for each patient | 10 years (01/01/2008-01/01/2018)
Date of death if occured | 10 years (01/01/2008-01/01/2018)
Cause of death | 10 years (01/01/2008-01/01/2018)
  Secondary to leukemia, treatment or other cause